CLINICAL TRIAL: NCT01259700
Title: China Rural Health Initiative: High Cardiovascular Risk Management and Salt Reduction in Rural Villages in China -- Two Parallel Large Cluster Randomized Controlled Trials
Brief Title: High Cardiovascular Risk Management and Salt Reduction in Rural Villages in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00025963; HHSN268200900027C (Other Grant/Funding Number: US NIH NHLBI (BAA contract))
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Disease
Keywords: High blood pressure; Primary care; Cardiovascular disease prevention; Salt reduction
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High risk management (Experimental)
  Interventions: Behavioral: High-risk patient standardized management package
- Salt reduction (Experimental)
  Interventions: Behavioral: Community based salt reduction program
- high risk management and salt reduction (Experimental)
  Interventions: Behavioral: High-risk patient standardized management package; Behavioral: Community based salt reduction program
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: High-risk patient standardized management package — A primary-care based high cardiovascular risk management package delivered by village doctors
  Other Names: high risk management
  Arms: High risk management; high risk management and salt reduction
Behavioral: Community based salt reduction program — A community-based salt reduction program delivered mainly by community health educators
  Other Names: Salt reduction
  Arms: Salt reduction; high risk management and salt reduction

SUMMARY:
Cardiovascular disease is the leading cause of death in China. At the village level, strategies for the control of cardiovascular disease are mostly absent. National clinical guidelines for the management of hypertension and cardiovascular disease are rarely disseminated to, or implemented by, the village primary care providers. Salt reduction has greater potential in rural China than almost anywhere else in the world. Very high levels of salt consumption, very little use of processed food and most dietary salt deriving from home cooking makes the removal of salt from the diet easier, cheaper and more worthwhile than in almost any other setting. The two large-scale cluster-randomized controlled trials proposed here will precisely and reliably define the effect of two highly plausible intervention strategies on important clinical outcomes. The evidence provided by the project will form the basis for policy setting that has the potential to greatly reduce the occurrence of vascular disease in rural China and take an important step towards balancing the rural urban divide in health and healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed history of coronary heart disease, ischemic stroke, or hemorrhagic stroke, or
* Older age (50 years or older for men; 60 years or older for women) and having physician-diagnosed Type I or Type II diabetes
* Older age (50 years or older for men; 60 years or older for women) and systolic blood pressure 160 mmHg (note that for simplicity, diastolic blood pressure is not included in the criteria)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mean systematic blood pressure level | October 2010 - December 2012
24 hour urinary sodium | October -December 2012

SECONDARY OUTCOMES:
24 hour urinary potassium | October-December 2012
Urinary sodium:potassium ratio | October-December 2012
Receiving regular primary care | October 2010 -December 2012
Taking anti-hypertensive medications | October 2010 -December 2012
Taking aspirin | October 2010 -December 2012
Receiving therapeutic lifestyle recommendations from village doctors | Oct 2010 - Dec 2012

OTHER OUTCOMES:
Knowledge, attitude and behaviour relating to salt consumption | October-December 2012
Awareness, treatment, and control of hypertension | October 2010 - December 2012

CONTACTS AND LOCATIONS:
Overall Officials: Yangfeng Wu, PhD, Principal Investigator — The George Institute for Global Health, China
Locations (5):
- China (5):
  - Hebei Province Center for Disease Prevention and Control ,China, Shijiazhuang, Hebei
  - The First Hospital Of China Medical University, Shenyang, Liaoning
  - Ningxia Medical University School of Public Health, Yinchuan, Ningxia
  - Changzhi Medical College, China, Changzhi, Shanxi
  - The Xi'an Jiaotong University School of Public Health, Xi’an, Shanxi

REFERENCES:
- [Derived] Chen S, Yan LL, Feng X, Zhang J, Zhang Y, Zhang R, Zhou B, Wu Y. Population-wide impact of a pragmatic program to identify and manage individuals at high-risk of cardiovascular disease: a cluster randomized trial in 120 villages from Northern China. Front Cardiovasc Med. 2024 May 24;11:1372298. doi: 10.3389/fcvm.2024.1372298. eCollection 2024. PMID 38854653
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803
- [Derived] Jardine MJ, Li N, Ninomiya T, Feng X, Zhang J, Shi J, Zhang Y, Zhang R, Zhang J, Hao J, Perkovic V, Heerspink HL, Wu Y, Yan LL, Neal B. Dietary Sodium Reduction Reduces Albuminuria: A Cluster Randomized Trial. J Ren Nutr. 2019 Jul;29(4):276-284. doi: 10.1053/j.jrn.2018.10.009. Epub 2018 Dec 24. PMID 30591358
- [Derived] Li N, Yan LL, Niu W, Yao C, Feng X, Zhang J, Shi J, Zhang Y, Zhang R, Hao Z, Chu H, Zhang J, Li X, Pan J, Li Z, Sun J, Zhou B, Zhao Y, Yu Y, Engelgau M, Labarthe D, Ma J, MacMahon S, Elliott P, Wu Y, Neal B. The Effects of a Community-Based Sodium Reduction Program in Rural China - A Cluster-Randomized Trial. PLoS One. 2016 Dec 9;11(12):e0166620. doi: 10.1371/journal.pone.0166620. eCollection 2016. PMID 27935977
- [Derived] Wang X, Li X, Vaartjes I, Neal B, Bots ML, Hoes AW, Wu Y. Does education level affect the efficacy of a community based salt reduction program? - A post-hoc analysis of the China Rural Health Initiative Sodium Reduction Study (CRHI-SRS). BMC Public Health. 2016 Aug 11;16(1):759. doi: 10.1186/s12889-016-3454-6. PMID 27515930
- [Derived] Zhang J, Wu T, Chu H, Feng X, Shi J, Zhang R, Zhang Y, Zhang J, Li N, Yan L, Niu W, Wu Y. Salt intake belief, knowledge, and behavior: a cross-sectional study of older rural Chinese adults. Medicine (Baltimore). 2016 Aug;95(31):e4404. doi: 10.1097/MD.0000000000004404. PMID 27495056
- [Derived] Yan LL, Fang W, Delong E, Neal B, Peterson ED, Huang Y, Sun N, Yao C, Li X, MacMahon S, Wu Y. Population impact of a high cardiovascular risk management program delivered by village doctors in rural China: design and rationale of a large, cluster-randomized controlled trial. BMC Public Health. 2014 Apr 11;14:345. doi: 10.1186/1471-2458-14-345. PMID 24721435